CLINICAL TRIAL: NCT03804983
Title: Safety and Efficacy of Initializing the Control-IQ Artificial Pancreas System Using Total Daily Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Tandem Diabetes Care, Inc. (Industry); DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Marc Breton, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 180030
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Artificial Pancreas (AP); Insulin Pump; Continuous Glucose Monitor (CGM); MyTDI; Hybrid Closed Loop (HCL); Total Daily Insulin (TDI)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: This trial aims to demonstrate the safety and feasibility of using MyTDI to determine insulin parameters on the Closed Loop Control (CLC) Artificial Pancreas (AP) System t:slim X2 with Control-IQ technology for use both at ski camp and at home in adolescent patients with type 1 diabetes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Hybrid Closed Loop (HCL) (Active Comparator): Eligible participants will be screened and enter the data collection period for approximately 5 days at home. Prior to participating in the 72-hour ski admission, participants will be randomized 1:1 to the use of Control-IQ with Hybrid Closed Loop (HCL) or the Control-IQ with MyTDI. Participants randomized to Control-IQ, participants will continue using their home insulin parameters during the ski admission and then 5 additional days at home.
  Interventions: Device: Hybrid Closed Loop (HCL)
- Control-IQ with MyTDI (Experimental): Eligible participants will be screened and enter the data collection period for approximately 5 days at home. Prior to participating in the 72-hour ski admission, participants will be randomized 1:1 to the use of Control-IQ or the Control-IQ with MyTDI. Participants randomized to Control-IQ with MyTDI, participants will be adjusted as noted below during the ski admission and will then continue these parameters for 5 additional days at home:
  * A single basal rate equal to total daily insulin (TDI)/48 will be implemented across the whole day
  * A single correction factor (CF) of 1650/TDI will be implemented across the whole day
  * Carbohydrate ratios (CR) will be set at:
    * 00:00-04:00 CR=450/TDI
    * 04:00-11:00 CR=360/TDI
    * 11:00-00:00 CR=450/TDI TDI will be set at the internal Control-IQ estimation total daily dose; if not available, total daily dose over the last 5 days will be used.
  Interventions: Device: Control-IQ with MyTDI

INTERVENTIONS:
Device: Hybrid Closed Loop (HCL) — Participants will use Control-IQ with Hybrid Closed Loop (HCL) with their own insulin parameters during the entire two-week study, including the 72-hour ski admission and the at-home study collection times. Parameters will be reduced 20% during the ski admission to adjust for the increased activity.
  Arms: Hybrid Closed Loop (HCL)
Device: Control-IQ with MyTDI — Participants will use their own insulin parameters during the first 5 days of the study. After randomization at the ski admission, the participants insulin parameters will be modified using the MyTDI calculations. Additionally, parameters will be reduced 20% during the ski admission to adjust for the increased activity.
  Arms: Control-IQ with MyTDI

SUMMARY:
The purpose of this proposed study is to assess the use of a new feature of the Control-IQ system, MyTDI.

DETAILED DESCRIPTION:
This trial aims to demonstrate the safety and feasibility of using MyTDI to determine insulin parameters on the Closed Loop Control (CLC) Artificial Pancreas (AP) system t:slim X2 with Control-IQ technology for use both at ski camp and at home in adolescent patients with type 1 diabetes.

Once deemed eligible, participants and their parent(s) will be trained on the use of the Tandem t:slim X2 insulin pump with Control-IQ technology and the study Dexcom G6 system. Participants will then use the this study equipment with their home insulin parameters at home for at home for 5 days. Participants will then come to the ski resort to participate in a 72-hour ski admission. Upon arrival, each participant will be randomized to either the using the Control-IQ system with their usual insulin parameters during the ski study and the at-home 5 days at home study or using the MyTDI insulin parameters during the ski study and the at-home 5 days at home study. Study duration for each participant will require 5 study visits over about 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for documented hyperglycemia (at least 1 must be met):

  * Clinical diagnosis of type 1 diabetes (C-peptide levels and antibody determinations are not required)
  * Diagnosis of type 1 diabetes is based on the investigator's judgement
* Criteria for requiring insulin at diagnosis (both criteria must be met):

  * Daily insulin therapy for ≥ 6 months
  * Insulin pump therapy for ≥ 3 months
* Age 12-18 years
* Currently using no insulins other than one of the following rapid-acting insulins at the time of enrollment: insulin lispro (Humalog), insulin aspart (Novolog), or insulin glulisine (Apidra). If using glulisine, subject must be willing to switch to lispro or aspart.
* Treatment with any non-insulin glucose-lowering agent (including GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, biguanides, sulfonylureas, and naturaceuticals) is permitted if stable on current dose for at least 1 month.
* Willingness to wear a continuous glucose sensor and physiological monitor for the duration of the study.
* For females, not pregnant or breastfeeding. Female subjects who are sexually active should agree to use birth control during the study.
* Total daily insulin dose (TDD) at least 10 U/day.

Exclusion Criteria:

* Diabetic ketoacidosis in the past 6 months
* Hypoglycemic seizure or loss of consciousness in the past 6 months
* History of seizure disorder
* History of any heart disease including coronary artery disease, heart failure, or arrhythmias
* History of altitude sickness
* Chronic pulmonary conditions that could impair oxygenation
* Cystic fibrosis
* Current use of oral glucocorticoids, beta-blockers or other medications, which in the judgement of the investigator, would be a contraindication to participation in the study.
* History of ongoing renal disease (other than microalbuminuria).
* Subjects requiring intermediate or long-acting insulin (such as NPH, Detemir, or Glargine).
* Pregnancy
* Presence of a febrile illness within 24 hours of the Ski Admission
* Medical or psychiatric conditions that in the judgement of the investigator might interfere with the completion of the protocol such as:

  * Inpatient psychiatric treatment in the past 6 months
  * Uncontrolled adrenal insufficiency
  * Alcohol abuse

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc D. Breton, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals within the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available after the primary publications of each study.
Access Criteria: Complete data sets will be provided to industry partners who would use the data for regulatory clearance (PMA - pre-market approval) of the tested artificial pancreas system. This will be done in response to the specific requirements of RFA-DK-14-024 for this project to "…generate data able to satisfy safety and efficacy requirements by regulatory agencies regarding the clinical testing of artificial pancreas device systems" in the target population of people with type 1 diabetes.

REFERENCES:
- [Background] Schoelwer MJ, Robic JL, Gautier T, Fabris C, Carr K, Clancy-Oliveri M, Brown SA, Anderson SM, DeBoer MD, Chernavvsky DR, Breton MD. Safety and Efficacy of Initializing the Control-IQ Artificial Pancreas System Based on Total Daily Insulin in Adolescents with Type 1 Diabetes. Diabetes Technol Ther. 2020 Aug;22(8):594-601. doi: 10.1089/dia.2019.0471. Epub 2020 Mar 2. PMID 32119790

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 22 enrolled participants, 20 were randomized to treatment. One participant was dropped after meeting stopping criteria.
Pre-assignment Details: 1 participant dropped prior to randomization for personal reasons (travel issues); 1 participant dropped prior to randomization as they didn't attend screening appointment.
Groups:
- Control-IQ With MyTDI: Eligible participants will be screened and enter the data collection period for approximately 5 days at home. Prior to participating in the 72-hour ski admission, participants will be randomized 1:1 to the use of Control-IQ or the Control-IQ with MyTDI. Participants randomized to Control-IQ with MyTDI, participants will be adjusted as noted below during the ski admission and will then continue these parameters for 5 additional days at home:
  * A single basal rate equal to total daily insulin (TDI)/48 will be implemented across the whole day
  * A single correction factor (CF) of 1650/TDI will be implemented across the whole day
  * Carbohydrate ratios (CR) will be set at:
    * 00:00-04:00 CR=450/TDI
    * 04:00-11:00 CR=360/TDI
    * 11:00-00:00 CR=450/TDI TDI will be set at the internal Control-IQ estimation total daily dose; if not available, total daily dose over the last 5 days will be used.
  Control-IQ with MyTDI: Participants will use their own insulin parameters during the first 5 days of the study. After randomization at the ski admission, the participants insulin parameters will be modified using the MyTDI calculations. Additionally, parameters will be reduced 20% during the ski admission to adjust for the increased activity.
Period: Overall Study
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Family Obligation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 10 | 20
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (1.7) | 14.7 (1.6) | 14.5 (1.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Time in Range at Home Pre/Post Intervention at Home
Description: The primary outcome for this study is the percent of time spent between 70mg/dL and 180mg/dL as computed by the number of CGM values falling in this interval divided by the total number of available CGM values. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Mean (Standard Deviation); unit: percentage of time spent in range
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage of time spent in range
  Baseline | 77.8 (6.2) | 70.7 (12.4)
  Home | 68.9 (8.9) | 70.1 (14.4)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.178, ANOVA — All outcomes were analyzed using repeated measure ANOVA comparing baseline to the studied period(i.e., ski admission or home use), grouped by treatment. Significance level was set at a P-Value<0.05

2. Secondary Outcome: Average CGM at Home
Description: Average of available CGM values within time frame
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
mg/dL
  Baseline | 142.4 (13.6) | 152.2 (19.2)
  Week 2-Home Portion | 156.5 (14.9) | 152.9 (21.2)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.145, ANOVA — [p-value comment as in outcome 1, analysis 1]

3. Secondary Outcome: Average CGM at Camp
Description: average of CGM values within time frame
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
mg/dL
  Baseline | 142.4 (13.6) | 152.2 (19.2)
  Camp | 144.3 (24.6) | 141.3 (13.1)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.304, ANOVA — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of CGM Values Below 50mg/dL at Home
Description: the percentage of CGM values falling below 50mg/dL, calculated as the number of CGM values <50mg/dL within the time frame divided by the total number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.0 [0.0 to 0.3] | 0.0 [0.0 to 0.1]
  Home | 0.0 [0.0 to 0.1] | 0.6 [0.0 to 0.8]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.131, ANOVA — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of CGM Values Below 50mg/dL at Camp
Description: the percentage of CGM values falling below 50mg/dL, computed as the number of CGM values <50mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (Baseline)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.0 (0.0) | 0.0 (0.0)
  Camp | 0.3 (0.7) | 0.16 (0.36)

6. Secondary Outcome: Percentage of CGM Values Below 54mg/dL at Camp
Description: the percentage of CGM values falling below 54mg/dL. computed as the number of CGM values <54mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.1 [0.0 to 0.6] | 0.1 [0.0 to 0.3]
  Camp | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.7]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.206, ANOVA — [p-value comment as in outcome 1, analysis 1]

7. Secondary Outcome: Percentage of CGM Values Below 60mg/dL at Home
Description: the percentage of CGM values falling below 60mg/dL. computed as the number of CGM values <60mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.7 [0.2 to 1.1] | 0.7 [0.0 to 0.8]
  Home | 0.5 [0.0 to 0.6] | 1.3 [0.1 to 1.8]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.335, ANOVA — [p-value comment as in outcome 1, analysis 1]

8. Secondary Outcome: Percentage of CGM Values Below 60mg/dL at Camp
Description: as for outcome 7
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (Baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.7 [0.2 to 1.1] | 0.7 [0.0 to 0.8]
  Camp | 0.5 [0.0 to 0.5] | 0.9 [0.0 to 2.3]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.637, ANOVA — [p-value comment as in outcome 1, analysis 1]

9. Secondary Outcome: Percentage of CGM Values Below 70mg/dL at Home
Description: the percentage of CGM values falling below 70mg/dL, computed as the number of CGM values <70mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 1.9 [0.6 to 5.3] | 2.1 [0.7 to 3.2]
  Home | 0.9 [0.3 to 1.9] | 2.4 [0.7 to 3.7]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.347, ANOVA — [p-value comment as in outcome 1, analysis 1]

10. Secondary Outcome: Percentage of CGM Values Below 70mg/dL at Camp
Description: as for outcome 9
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (Baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 1.9 [0.6 to 5.3] | 2.1 [0.7 to 3.2]
  Camp | 1.4 [0.0 to 2.4] | 3.8 [0.5 to 4.7]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.057, ANOVA — [p-value comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of CGM Values Between 70mg/dL and 180mg/dL at Camp
Description: the percentage of CGM values falling between 70mg/dL and 180mg/dL, computed as the number of CGM values <=180mg/dL and >70mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 77.8 (6.2) | 70.7 (12.4)
  Camp Portion | 78.4 (12.8) | 76.5 (8.0)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.435, ANOVA — [p-value comment as in outcome 1, analysis 1]

12. Secondary Outcome: Percentage of CGM Values Above 180mg/dL at Home
Description: the percentage of CGM values falling above 180mg/dL, computed as the number of CGM values >180mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 18.9 (17.7) | 26.9 (12.7)
  Home | 29.1 (10.3) | 27.2 (14.4)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.135, ANOVA — [p-value comment as in outcome 1, analysis 1]

13. Secondary Outcome: Percentage of CGM Values Above 180mg/dL at Camp
Description: as for outcome 12
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 18.9 (7.7) | 26.9 (12.7)
  Camp | 20.1 (13.4) | 20.1 (7.3)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.271, ANOVA — [p-value comment as in outcome 1, analysis 1]

14. Secondary Outcome: Percentage of CGM Values Above 250mg/dL at Home
Description: the percentage of CGM values falling above 250mg/dL, computed as the number of CGM values >250mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 3.4 [2.7 to 4.2] | 6.5 [1.7 to 9.3]
  Home | 5.8 [4.2 to 7.3] | 3.8 [1.8 to 9.3]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 1.0, ANOVA — [p-value comment as in outcome 1, analysis 1]

15. Secondary Outcome: Percentage of CGM Values Above 250mg/dL at Camp
Description: as for outcome 14
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 16 (13.6) | 10 (11.4)
  Camp | 14.88 (12.36) | 8.04 (10.14)

16. Secondary Outcome: Percentage of CGM Values Above 300mg/dL at Home
Description: the percentage of CGM values falling above 300mg/dL, computed as the number of CGM values >300mg/dL within the time frame divided by the number of available CGM values within the time frame. CGM gaps inferior to 3 hours will be linearly interpolated.
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.3 [0.0 to 0.8] | 0.3 [0.0 to 2.2]
  Home | 0.7 [0.2 to 3.2] | 0.9 [0.0 to 2.7]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 1.0, ANOVA — [p-value comment as in outcome 1, analysis 1]

17. Secondary Outcome: Percentage of CGM Values Above 300mg/dL at Camp
Description: as for outcome 16
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
percentage
  Baseline | 0.3 [0.0 to 0.8] | 0.3 [0.0 to 2.2]
  Camp | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.294, ANOVA — [p-value comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change in Total Daily Insulin at Home
Description: sum of the recorded insulin injection over the time frame in units
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
Units
  Baseline | 39.0 (7.3) | 48.7 (18.4)
  Home | 48.2 (11.2) | 54.9 (29.0)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.584, ANOVA — [p-value comment as in outcome 1, analysis 1]

19. Secondary Outcome: Change in Total Daily Insulin at Camp
Description: sum of the recorded insulin injection over the time frame in units
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (baseline)
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
Units
  Baseline | 39.0 (7.3) | 48.7 (18.4)
  Camp | 38.8 (11.3) | 50.9 (27.5)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.69, ANOVA — [p-value comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change in Total Meal Carbohydrates at Home
Description: sum of the meal sized recorded over the time frame
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
Grams
  Baseline | 226.3 (38.6) | 204.1 (100.4)
  Home | 276.5 (94.5) | 192.6 (115.4)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.066, ANOVA — [p-value comment as in outcome 1, analysis 1]

21. Secondary Outcome: Change in Total Meal Carbohydrates at Camp
Description: sum of the meal sized recorded over the time frame
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (Baseline)
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
Grams
  Baseline | 226.3 (38.6) | 204.1 (100.4)
  Camp | 280.0 (43.0) | 254.6 (143.5)
Statistical Analysis 1: Comparison: Hybrid Closed Loop (HCL) vs Control-IQ With MyTDI; Test type: Other — Analysis of Variance; p = 0.904, ANOVA — [p-value comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change in Number of Hypoglycemic Events at Camp
Description: Sum of hypoglycemic events within the time frame. An event is defined by a group of consecutive CGM values below 70 mg/dL)
Time Frame: 2 days during camp admission (Camp) compared to 5 days prior to camp (Baseline)
Measure: Median (Inter-Quartile Range); unit: events per day
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
events per day
  Baseline | 1 [0.4 to 2] | 0.5 [0.4 to 1.4]
  Camp | 1 [0 to 1] | 1 [0.5 to 2.5]

23. Secondary Outcome: Number of Hypoglycemia Treatment at Camp
Description: Sum of the number of CHO treatments recorded over the time frame
Time Frame: 2 days during camp admission (Camp)
Measure: Median (Inter-Quartile Range); unit: events per day
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
events per day | 1.5 [1 to 2.5] | 2.5 [0 to 3]

24. Secondary Outcome: Total Amount of Carbohydrates Corresponding to Hypoglycemia Treatment at Camp
Description: Sum of the amount of carbohydrates used for treatments recorded over the time frame
Time Frame: 2 days during camp admission (Camp)
Measure: Mean (Standard Deviation); unit: grams per day
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
grams per day | 35.9 (37) | 43.6 (35.2)

25. Secondary Outcome: Change in Hypoglycemia Events at Home
Description: change in number of hypoglycemia between baseline and home
Time Frame: 5 days post camp (home) compared to 5 days before camp (baseline)
Measure: Median (Inter-Quartile Range); unit: events per day
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
Number analyzed (Participants) | 9 | 9
events per day
  Baseline | 1 [0.4 to 2] | 0.6 [0.4 to 1.4]
  Home | 0.3 [0.2 to 0.8] | 0.7 [0.2 to 1.3]

ADVERSE EVENTS:
Time Frame: 13 days
Description: Any untoward medical occurrence in a study participant, irrespective of the relationship between the adverse event and the device(s) under investigation
Arm/Group | Hybrid Closed Loop (HCL) | Control-IQ With MyTDI
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hybrid Closed Loop (HCL) (N=10) | Control-IQ With MyTDI (N=10)
Hyperglycemia or ketosis events without meeting criteria for Diabetes Ketoacidosis (Endocrine disorders) | 0 (0) | 1 (1)
Concussion (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory illness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT03804983/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03804983/ICF_001.pdf